CLINICAL TRIAL: NCT06147427
Title: ARAVET : Antero-lateral Ligament Reconstruction Versus Modified Lemaire's Lateral Extra-articular Tenodesis in Combination With ACL Reconstruction With a Minimum Follow up of 2 Years: a Randomized Controlled Trial
Brief Title: ALL Reconstruction Versus Modified Lemaire's LET in Combination With ACL Reconstruction With a Minimum Follow up of 2 Years
Acronym: ARAVET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL23_0851; id-rcb (Other: 2023-A02105-40)
Record Dates: First submitted 2023-11-17; First posted 2023-11-27 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: ACL reconstruction; lateral extra-articular tenodesis; modified Lemaire tenodesis; anterolateral ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL reconstruction with hamstrings combined with ALL plasty (Experimental): Patient treated by ACL reconstruction with hamstrings combined anterolateral plasty using the ALL reconstruction technique (Gracilis throught the femur tunnel of the ACL graft and fixed to the tibia by an anchor on its point of isometry on the tibia).
  Interventions: Procedure: ACL reconstruction with hamstrings combined with ALL plasty
- ACL reconstruction with hamstrings combined with modified Lemaire's LET (Experimental): Patient treated by ACL reconstruction with hamstrings combined with modified Lemaire's lateral extra-articular tenodesis technique (Fascia lata strip pedicled to the Gerdy and fixed to the femur throught the tunnel of the ACL graft).
  Interventions: Procedure: ACL reconstruction with hamstrings combined with modified Lemaire's LET

INTERVENTIONS:
Procedure: ACL reconstruction with hamstrings combined with ALL plasty — ACL reconstruction with hamstrings combined anterolateral plasty using the ALL reconstruction technique (Gracilis throught the femur tunnel of the ACL graft and fixed to the tibia by an anchor on its point of isometry on the tibia).
  Arms: ACL reconstruction with hamstrings combined with ALL plasty
Procedure: ACL reconstruction with hamstrings combined with modified Lemaire's LET — ACL reconstruction with hamstrings combined with modified Lemaire's lateral extra-articular tenodesis technique (Fascia lata strip pedicled to the Gerdy and fixed to the femur throught the tunnel of the ACL graft).
  Arms: ACL reconstruction with hamstrings combined with modified Lemaire's LET

SUMMARY:
Anterior cruciate ligament (ACL) tears are associated with concomitant lesions of the anterolateral ligament (ALL), which increase rotatory instability of the knee. If untreated, ALL insufficiency can compromise the results of ACL reconstruction, with higher risk of iterative ACL tear or additional meniscal lesion.

Several surgical techniques have been described to reconstruct the ALL. Indications are increasingly frequent and actually, consensus being young patients, patients practising pivot sports, significant rotational laxity on clinical examination with a positive pivot shift test, or in cases of iterative surgery. To date, the two most popular techniques are the Lemaire technique (use of a fascia lata strip) and LAL reconstruction plasty (use of part of an accessory hamstring tendon).

The older Lemaire procedure, popularized in the 1980s has proved its efficiency in terms of biomechanics, safety and reproducibility. More recently, following a new, precise anatomical description, anterolateral ligament plasty (ALL) has been developed, which is intended to be more anatomical than Lemaire's technique, but whose clinical superiority has not yet been demonstrated.

Both techniques are currently used in our department, with the choice of technique left to the surgeon's discretion.

To date, no randomized prospective study has demonstrated the clinical superiority of one technique over the other with a long term follow up.

The aim of this study was to compare graft survival of ALL reconstruction versus modified Lemaire LET in combination with ACL reconstruction with a minimum follow up of 2 years. Secondary aim was to compare functional outcomes between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman with age between 18 and 50 years old
* disabling anterior chronic laxity
* 1 criteria of anterolateral plasty indication : pivot sport, rotatory instability with positive pivot shift test
* Patient who signed the informed consent form.

Exclusion Criteria:

* any associated procedure (excluding meniscal resection or repair) like osteotomy or meniscus graft
* pregnant patient
* Persons deprived of their liberty by judicial or administrative decision, persons under psychiatric care
* Adults under legal protection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 248 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2029-01-16 (Estimated); Study Completion 2029-01-16 (Estimated)

PRIMARY OUTCOMES:
Graft rupture rate | At 24 months post-operative
  Graft rupture rate (percentage)

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) score | Pre-operatively and at 6, 12 and 24 months post-operatively
  Functional outcome : mean IKDC score
Complications | Pre-operatively and at Day 0, Day 21, Day 45, 6 months, 12 months and 24 months post-operatively
  Complications all causes

CONTACTS AND LOCATIONS:
Overall Officials: Elvire SERVIEN, MD, Principal Investigator — Service de chirurgie orthopédique et de médecine du sport
Locations (1):
- Service de chirurgie orthopédique et de médecine du sport, Lyon, France

IPD SHARING:
Plan to Share IPD: No